CLINICAL TRIAL: NCT02284750
Title: A Prospective, Multi-center, Randomized Trial Comparing Two-stent With Provisional Stenting Techniques for Patients With Complex Coronary Bifurcation Lesions
Brief Title: Two-stent vs Provisional Stenting Techniques for Patients With Complex Coronary Bifurcation Lesions
Acronym: DEFINITION-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NFH20141029
Record Dates: First submitted 2014-10-29; First posted 2014-11-06 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease
Keywords: Bifurcation lesion; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Two-stenting technique (Experimental): Percutaneous coronary intervention with DK crush, or culotte technique
  Interventions: Procedure: Percutaneous coronary intervention
- Provisional stenting technique (Active Comparator): Percutaneous coronary intervention with Provisional stenting technique. Stenting of the side branch was required if TIMI flow was <3, or ≥ type B dissection after kissing balloon inflation.
  Interventions: Procedure: Percutaneous coronary intervention

INTERVENTIONS:
Procedure: Percutaneous coronary intervention
  Other Names: PCI

SUMMARY:
The purpose of this study is to establish the optimal strategy for stenting in coronary bifurcation lesion.

DETAILED DESCRIPTION:
The current study is designed as a multicenter, randomized and prospective study aiming to compare the effect of two-stenting and simple stenting techniques in patients with complex bifurcation lesions. Based on the previous studies, the rate of 1-year target lesion failure events was around 14% after PCI with provisional stenting. And our previous data showed that this event at 12-month after two-stenting procedure was 7%. Considering the lost to follow-up, it is anticipated that up to 660 patients will be enrolled in the trial. All patients will have repeat angiography at 13 months, with clinical follow-up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures;
* Men and women 18 years and older;.
* Established indication to PCI according to the guidelines of American Heart Association and American College of Cardiology;
* Native coronary lesion suitable for drug-eluting stent placement;
* True bifurcation lesions (Medina 0,1,1/1,1,1);
* Reference vessel diameter in side branch ≥2.5mm by visual estimation;
* Complex bifurcation lesions based on DEFINITION study.

Exclusion Criteria:

* Pregnancy and breast feeding mother;
* Co-morbidity with an estimated life expectancy of < 50 % at 12 months;
* Scheduled major surgery in the next 12 months;
* Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk;
* Unable to provide written informed consent, or fail to follow the protocol;
* Previous enrolment in coronary intervention device investigation during the study period;
* Patient with STEMI within 24-hour from the onset of chest pain to admission;
* Restenosis bifurcation lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Target lesion failure | 12 months
  Combined end point of: cardiac death, target-vessel myocardial infarction (MI), or target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Cardiac death | 12 months
Target-vessel myocardial infarction | 12 months
Target lesion revascularisation | 12 months
Target vessel revascularisation | 12 months
Stent thrombosis | 12 months

OTHER OUTCOMES:
Acute gain | Intraoperative
  The acute gain was defined as the difference between post- and preprocedural minimal lumen diameter (MLD)
In-stent restenosis | 13 months
  In-stent restenosis was defined as ≥50% diameter stenosis at the follow-up angiogram.
Late lumen loss | 13 months
  The late lumen loss was defined as the difference between post- and follow-up minimal lumen diameter (MLD)

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kan J, Zhang JJ, Sheiban I, Santoso T, Munawar M, Tresukosol D, Xu K, Stone GW, Chen SL; DEFINITION II Investigators. 3-Year Outcomes After 2-Stent With Provisional Stenting for Complex Bifurcation Lesions Defined by DEFINITION Criteria. JACC Cardiovasc Interv. 2022 Jul 11;15(13):1310-1320. doi: 10.1016/j.jcin.2022.05.026. PMID 35798473
- [Derived] Zhang JJ, Ye F, Xu K, Kan J, Tao L, Santoso T, Munawar M, Tresukosol D, Li L, Sheiban I, Li F, Tian NL, Rodriguez AE, Paiboon C, Lavarra F, Lu S, Vichairuangthum K, Zeng H, Chen L, Zhang R, Ding S, Gao F, Jin Z, Hong L, Ma L, Wen S, Wu X, Yang S, Yin WH, Zhang J, Wang Y, Zheng Y, Zhou L, Zhou L, Zhu Y, Xu T, Wang X, Qu H, Tian Y, Lin S, Liu L, Lu Q, Li Q, Li B, Jiang Q, Han L, Gan G, Yu M, Pan D, Shang Z, Zhao Y, Liu Z, Yuan Y, Chen C, Stone GW, Han Y, Chen SL. Multicentre, randomized comparison of two-stent and provisional stenting techniques in patients with complex coronary bifurcation lesions: the DEFINITION II trial. Eur Heart J. 2020 Jul 14;41(27):2523-2536. doi: 10.1093/eurheartj/ehaa543. PMID 32588060
- [Derived] Zhang JJ, Gao XF, Han YL, Kan J, Tao L, Ge Z, Tresukosol D, Lu S, Ma LK, Li F, Yang S, Zhang J, Munawar M, Li L, Zhang RY, Zeng HS, Santoso T, Xie P, Jin ZN, Han L, Yin WH, Qian XS, Li QH, Hong L, Paiboon C, Wang Y, Liu LJ, Zhou L, Wu XM, Wen SY, Lu QH, Yuan JQ, Chen LL, Lavarra F, Rodriguez AE, Zhou LM, Ding SQ, Vichairuangthum K, Zhu YS, Yu MY, Chen C, Sheiban I, Xia Y, Tian YL, Shang ZL, Jiang Q, Zhen YH, Wang X, Ye F, Tian NL, Lin S, Liu ZZ, Chen SL. Treatment effects of systematic two-stent and provisional stenting techniques in patients with complex coronary bifurcation lesions: rationale and design of a prospective, randomised and multicentre DEFINITION II trial. BMJ Open. 2018 Mar 6;8(3):e020019. doi: 10.1136/bmjopen-2017-020019. PMID 29511018